CLINICAL TRIAL: NCT05087407
Title: Cutting Seton Versus Decompression and Drainage Seton in the Treatment of High Complex Anal Fistula
Brief Title: Decompression and Drainage Seton in the Treatment of High Complex Anal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hui Li, Associate chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.2016-81
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: High Complex Anal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- decomprssion and drainage seton (Experimental)
  Interventions: Procedure: Decomprssion and drainage seton
- Cutting seton (Active Comparator)
  Interventions: Procedure: Cutting seton

INTERVENTIONS:
Procedure: Decomprssion and drainage seton — Incision the internal sphincter over the fistula tract in intersphinteric space to achieve decompression then drainage seton will be put around external sphincter.
  Arms: decomprssion and drainage seton
Procedure: Cutting seton — Cutting seton is introduced from outside openning to internal openning and encircling the internal and external anal sphincter.
  Arms: Cutting seton

SUMMARY:
This study aimed to compare the efficacy of the decompression and drainage seton (DADS) and cutting seton (CS) in the treatment of high complex anal fistula.

ELIGIBILITY:
Inclusion Criteria:

* high trans-sphincteric cryptoglandular anal fistulas (involving >30% of the EAS muscles evaluated through magnetic resonance imaging (MRI) scan, endoanal ultrasonography)
* suprasphincteric fistulas were enrolled

Exclusion Criteria:

* Low anal fistula; -Non-glandular anal fistulas, such as tuberculous anal fistula and Crohn's anal fistula; -
* Patients with symptoms of fecal incontinence;
* A previous history of anal fistula surgical treatment;
* Patients with malignant tumors or mental illness or other reasons unable to cooperate with the treatment.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of healing | 6 months post-operation.
  complete healing was defined as complete epithelialization of the wound, with no evidence of external fistula opening or perianal discharge under physical examination.
Recurrence rate | within 12 months after the procedure
  recurrence was defined as the clinical reappearance of the fistula after complete healing, removal or fall-off of seton
The healing time of the anal wound (days) | 6 months post-operation.
  the time needed to achieve complete healing of anal fistula.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No